CLINICAL TRIAL: NCT02784522
Title: Minimally Invasive Treatment of Proximal Humerus Fractures With Locking Compression Plate Improves Shoulder Function in Older Patients: Study Protocol for a Prospective Randomized Controlled Trial
Brief Title: Minimally Invasive of Proximal Humerus Fractures With Internal Fixation Improves Shoulder Function in Older Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qinghai University (Other)
Responsible Party: Principal Investigator, Tao Wu, Director, Qinghai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QinghaiUH_001
Record Dates: First submitted 2016-05-19; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Humerus Fractures
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- locking compression plate group (Experimental): In the experimental group, patients will undergo closed reduction via a lateral approach to the shoulder followed by locking compression plate fixation using a minimally invasive technique.The locking compression plate is purchased from Xiamen Dabo Yingjing Medical Devices Co., Ltd., Xiamen, China.
  Interventions: Device: locking compression plate group
- conventional locking plate group (Active Comparator): Patients in the control group will be subjected to closed reduction via a lateral approach to the shoulder followed by conventional steel plate fixation using a minimally invasive technique. The conventional locking plate is purchased from Xiamen Dabo Yingjing Medical Devices Co., Ltd., Xiamen, China.
  Interventions: Device: conventional locking plate group

INTERVENTIONS:
Device: locking compression plate group — Closed reduction via shoulder lateral approach followed by locking compression plate fixation using minimally invasive technique
  Arms: locking compression plate group
Device: conventional locking plate group — Closed reduction via shoulder lateral approach followed by conventional locking plate fixation using minimally invasive technique
  Arms: conventional locking plate group

SUMMARY:
This study protocol represents an attempt to objectively choose appropriate methods for internal fixation of proximal humerus fractures in older patients by comparing locking compression plate with conventional steel plate fixation to improve shoulder function.

DETAILED DESCRIPTION:
Treatment for proximal humerus fractures emphasizes the restoration of shoulder function. Older patients, because of the loss of bodily functions, face enormous difficulties in fracture healing and shoulder functional recovery after sustaining proximal humerus fractures. As previously reported, open reduction with conventional locking plate fixation achieved fair outcomes in 48 cases of proximal humerus fractures in older patients, with an excellent rate of 85.4% according to the Neer classification system. The investigators' clinical experience, however, has shown that the stability of internal fixation is inadequate and must be enhanced. Consequently, the investigators design a microsurgical implantation using a locking compression plate (LCP) to treat proximal humerus fractures in older patients.

In a search of the Web of Science database, the investigators found a randomized controlled trial reported by Wang et al. in which LCP fixation using microsurgical techniques had better outcomes in 20 cases of proximal humerus fractures in older patients. However, the limitation created by the small sample size had profound effects on the reliability of their study.

No relevant articles were retrieved from the Chinese Clinical Trial Register, and only one similar article was found on ClinicalTrials.gov: "Proximal Humerus Fractures: Randomized Study Between Locking Nails and Locking Plates for Neer 2 and 3 Parts" (identifier: NCT01984112). In this clinical trial, Constant-Murley scores were considered the primary outcome, and the follow-up period was 12 months. Importantly, the inclusion criteria and study arms were distinctly different from those in the investigators' study protocol.

The main principle of minimally invasive techniques in orthopedics is to implant a specific bony plate, which is fixed across a transverse fracture, via small incisions of the periosteum, skin, and muscle. These implantation devices include less invasive stabilization systems, dynamic compression plate systems, and LCP systems. Internal fixation with the LCP system involves two completely different fixation techniques and two opposing osteosynthesis principles, namely conventional plate and bridging plate osteosyntheses characterized by direct anatomical reduction. Because of its special design, the LCP can be used as a dynamic compression plate, as a pure internal fixator using locking head screws, or as both combined, thus providing a variety of therapeutic options for surgeons. Moreover, the LCP has good stability and induces less damage to the periosteum; it is therefore beneficial for bone healing and functional recovery. Given these characteristics, the LCP is likely to have stronger stability than the conventional locking plate for internal fixation of fractures. Therefore, the investigators design a study protocol that compares the LCP and conventional locking plate using minimally invasive techniques for internal fixation of proximal humerus fractures in older patients. The investigators hypothesize that the LCP will be more effective than the conventional locking plate in promoting shoulder function recovery with a higher excellent rate according to the Neer classification system for proximal humerus fractures.

Data collection, management, analysis, and open access

* Data collection: All data, including demographic information, disease diagnosis, concomitant diseases, allergic history (drug allergy), and adverse reactions, will be collected on a case report form and summarized in one form. These data will be recorded electronically using a double-data entry strategy by EpiData software.
* Data management: Only the project manager will have the right to query the database, and changes will not be allowed. All data relevant to this clinical trial will be preserved by the Affiliated Hospital of Qinghai University.
* Data analysis: All data will be statistically analyzed by professional statisticians. The statistical report by the statisticians will be given to the project manager responsible for writing the research report. An independent data monitoring committee will be in charge of data monitoring and management throughout the entire trial to ensure scientific accuracy, authenticity, and integrity.
* Open data: Published data will be released at www.figshare.com.

Statistical analysis The statistical analysis will be completed by statisticians using the SPSS 19.0 statistical software (IBM Corp., Armonk, NY, USA) in line with the intention-to-treat principle. Intergroup comparison for the excellent rate according to the Neer classification system will be performed using the chi-square test. The operation time, intraoperative blood loss, postoperative hospital stay, fracture healing time, visual analogue scale scores, and SF-36 scores will be compared using the Mann-Whitney U test. A value of P < 0.05 will be considered statistically significant.

Adverse events

* Predicted and unanticipated adverse events will be recorded during the trial.
* Adverse events including dizziness, fever, infection, subacromial impingement, humeral head necrosis, malunion, and severe pain will be detected.
* All serious adverse events will be recorded in detail, including the date of occurrence, type of event, and treatments, all of which will be reported to the project manager and institution review board within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Neer II or III fractures as shown by X-ray examination
* Presentation with soft tissue swelling of the shoulder, limited mobility, tenderness, unusual activity, or a palpable sense of bone rubbing
* Unilateral traumatic fracture
* Over 60 years of age
* Admission to the hospital within 6 hours after injury
* Informed consent from patients or their relatives

Exclusion Criteria:

* Concomitant injuries involving pathological fracture, blood vessel injury, or nerve injury
* Head-split humerus fractures
* Severe comminuted proximal humerus fractures involving > 40% of the articular surface of the humeral head
* Disturbance of consciousness, cerebral infarction, cancer, severe medical complications (such as heart, lung, or kidney failure; severe hypertension; diabetes; or blood diseases)
* History of shoulder or elbow dysfunction

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Neer classification system score | month 6 after surgery
  Clinical outcome scores according to the Neer classification system will be used to assess shoulder function recovery.

SECONDARY OUTCOMES:
change of visual analogue scale score | day 1, day 3 and week 1, week 2 after surgery
  Visual analogue scale scores assess postoperative pain relief.
change of X-ray examinations | month 0.5, month 1, month 3, and month 6 after surgery
  Disappearance of the fracture line shown on X-ray examination indicates fracture healing.
Change of Medical Outcomes Study 36-item Short Form Health Survey (SF-36) Score | month 0.5, month 1, month 3, and month 6 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wu, Master, Principal Investigator — Affiliated Hospital of Qinghai University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196